CLINICAL TRIAL: NCT01058629
Title: A 180 Day, Multicenter Study to Evaluate the Clinical Performance of SynergEyes A2 Hybrid Contact Lenses for Daily Wear Use in the Correction of Refractive Error With or Without Astigmatism in Non-diseased Eyes
Brief Title: Study to Evaluate the Clinical Performance of SynergEyes A2 Hybrid Contact Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SynergEyes, Inc. (Industry)
Responsible Party: Jennifer Callahan, MAS/Manager of Clinical and Regulatory Affairs, SynergEyes, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI 09-01
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Refractive Errors; Astigmatism
Keywords: Hybrid; contact lens; myopia; hyperopia; near sighted; astigmatism; far sighted
MeSH Terms: conditions — Refractive Errors; Astigmatism; Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SynergEyes A2 Hybrid Contact Lens (Experimental)
  Interventions: Device: SynergEyes A2 Hybrid Contact Lens

INTERVENTIONS:
Device: SynergEyes A2 Hybrid Contact Lens — SynergEyes A2 is a hybrid contact lens cleared by the US Food and Drug Administration (FDA) for daily wear correction of up to +20.00 and -20.00 in eyes with astigmatism up to 6.00D and for presbyopia.

SUMMARY:
This is a multicenter study to evaluate the clinical performance of the SynergEyes A2 lens in patients with refractive errors with or without astigmatism.

DETAILED DESCRIPTION:
Hybrid contact lenses have been previously shown to be a safe and effective method to correct refractive errors with and without astigmatism. The hybrid contact lens design may provide greater visual acuity and comfort than other soft or rigid gas permeable (RGP) lenses currently available. The purpose of this study is to confirm the design of the SynergEyes A2 lens by evaluating clinical performance and, if necessary, modify certain lens parameters in order to optimize lens performance. Objective and subjective parameters will be used to evaluate the lens.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand and be willing to sign a written informed consent form
* Age ≥18 years
* Be willing and able to adhere to the instructions set forth in this protocol and able to keep all specific appointments
* Have naturally occurring myopia up to -6.00 D or hyperopia up to +2.00 D (spectacle plane) with or without corneal astigmatism up to 6.00 D
* Be in good general health, based on his/her knowledge, including normal healthy eyes
* Possess wearable and visually functional eyeglasses
* Have manifest refraction visual acuity equal to or better than 20/25 in each eye

Exclusion Criteria:

* Subject requires multifocal vision correction or is wearing lenses in a monovision modality
* Subject has lenticular astigmatism uncorrectable by normal RGP tear layer optics
* Subject exhibits poor personal hygiene
* Subject is currently or within 30 days prior to enrollment in this study has been an active participant in another clinical study (except SynergEyes Protocol # SI 08-05)
* Subject is currently pregnant (to the best of the subject's knowledge), is planning a pregnancy within the next 9 months, or is lactating
* Subject has a known sensitivity to ingredients used in contact lens care products
* Subject has undergone refractive surgery or is currently receiving or has previously received orthokeratology treatment
* Subject is aphakic or pseudophakic
* Subject has ocular or systemic disease such as, but not limited to, anterior uveitis or iritis (past or present), glaucoma, Sjogren's Syndrome, lupus erythematosus, scleroderma, keratoconus, post surgical corneal irregularity or type II diabetes
* Subject is using ocular medications for any reason or systemic medications which might interfere with contact lens wear
* A known history of corneal hypoesthesia (reduced corneal sensitivity)
* Slit lamp findings that would contraindicate contact lens wear, including, but not limited to:

  * Evidence of corneal ulcer, corneal infiltrates or fungal infections
  * Corneal scars within the visual axis
  * Pterygium
  * Dry eye symptoms with decrease tear levels and punctuate staining ≥ Grade 2
  * Neovascularization or ghost vessels ≥1.5mm in from the limbus
  * Seborrhoeic eczema or seborrhoeic conjunctivitis
  * History of papillary conjunctivitis that has interfered with lens wear or a current condition of Grade 2 or greater
* Clinically significant (Grade 3 or 4) anterior segment abnormalities or any infection of the eye, lids or associated structures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Confirm current SynergEyes A2 lens design by evaluating clinical performance using objective and subjective parameters | 6 months

SECONDARY OUTCOMES:
Determine the best method for fitting the SynergEyes A2 hybrid contact lens | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kusy, OD, MS, FAAO, Principal Investigator — SynergEyes, Inc.
Locations (10):
- United States (10):
  - Family Eye Care Center, Campbell, California
  - SynergEyes, Inc., Carlsbad, California
  - Encino Optometric Center Corp., Encino, California
  - Carmel Mountain Vision Care, San Diego, California
  - VisionCare Associates, PC, East Lansing, Michigan
  - The Koetting Associates, St Louis, Missouri
  - Eyesite, Penfield, New York
  - Primary Eyecare Group, Brentwood, Tennessee
  - Specialty Eyecare Group Totem Lake Vision Center, Kirkland, Washington
  - Snowy Range Vision Center, Laramie, Wyoming